CLINICAL TRIAL: NCT03652506
Title: Investigation the Effect of Regional Anesthesia Methods Anterior Abdominal Wall Tissue Oxygenation on Laparoscopic Cholecystectomy
Brief Title: The Impact of Anterior Abdominal Wall Tissue Oxygenation During Pneumoperitoneum of Regional Anesthesia Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2018/06-27
Record Dates: First submitted 2018-08-19; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Laparoscopy; Abdominal Wall; Regional Anesthesia

STUDY DESIGN:
Intervention Model Description: prospective,randomized
Who Masked: Participant
Masking Description: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Interventions: Device: regional oxymetry probe
- Group E (Active Comparator): Thoracic Epidural block +The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Interventions: Device: regional oxymetry probe; Procedure: Thoracic Epidural block
- Group Q (Active Comparator): Ultrasound guided unilateral anterior Quadratus Lumborum block +The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Interventions: Device: regional oxymetry probe; Procedure: Quadratus Lumborum block

INTERVENTIONS:
Device: regional oxymetry probe — The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Other Names: abdominal wall tissue oxygenation
Procedure: Quadratus Lumborum block — Ultrasound guided unilateral anterior Quadratus Lumborum block with 20 ml %0.25 bupivacaine+The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Arms: Group Q
Procedure: Thoracic Epidural block — Thoracic Epidural block with 20 ml %0.25 bupivacaine+The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Arms: Group E

SUMMARY:
During laparoscopic surgery, the abdomen is inflated with carbon dioxide for abdominal imaging and increased intraabdominal pressure affects intraabdominal structures and abdominal wall.

DETAILED DESCRIPTION:
The investigators aimed to investigate the effects of regional anesthesia methods administered during laparoscopic cholecystectomy on abdominal wall oxygenation and postoperative pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class
* Underwent laparoscopic cholecystectomy

Exclusion Criteria:

* Previous surgeon surgeon
* Local anesthetic allergy,
* Bleeding is a diathesis disorder
* Mental impairment,
* Allergic to the drugs used,
* Patients who are not reluctant to participate in the study,
* Presence of infection in the block area,
* Patients whose body mass index is over 30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-28 (Estimated); Primary Completion 2018-12-28 (Estimated); Study Completion 2018-12-28 (Estimated)

PRIMARY OUTCOMES:
rso2 | peroperative 2 hours
  The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line

SECONDARY OUTCOMES:
Visual Analog Scale | Postoperative 24 hours
  Visual Analog Scale was used for pain.Pain intensity was measured using 0-10 cm visual analogue scale (VAS). (0=no pain, 10=intolerable pain)
tramadol consumption | Postoperative 24 hours
  tramadol consumption with PCA (patient-controlled analgesia ) device
additional analgesic use | Postoperative 24 hours
  additional analgesic use (paracetamol and NSAİD)

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, M.D, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No